CLINICAL TRIAL: NCT01739114
Title: Sustained Inflations to Achieve Lung Aeration at Birth - a Randomized Control Trial
Brief Title: Assessment of Lung Aeration at Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Georg Schmolzer, Research Neonatologist, Postdoctoral Fellow, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00034524
Record Dates: First submitted 2012-11-27; First posted 2012-12-03 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Lung aeration; Bronchopulmonary dysplasia; Positive Pressure Respiration; Sustained Inflation; Continuous Positive Airway Pressure
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "SI group" (Experimental): Infants randomized into the "SI group" will receive two initial sustained inflations with a PIP of 20 cm H2O.
  After the two initial SIs infants will receive PEEP of 5 cm H2O and then CPAP if breathing spontaneously or, if found to have apnea or laboured breathing, mask IPPV with a PIP of 20 cm H2O and PEEP of 5 cm H2O at a rate of 40 to 60 bpm until spontaneously breathing, at which time CPAP will be provided.
  Interventions: Procedure: SI group
- IPPV group (Active Comparator): Infants randomized into the "IPPV group" will receive mask IPPV with an initial PIP of 20 cmH2O and PEEP of 5 cm H2O, and a ventilation rate of 40-60 inflations/min until spontaneously breathing, at which time CPAP will be provided.
  Interventions: Procedure: "IPPV group"

INTERVENTIONS:
Procedure: "IPPV group" — Infants randomized into the "IPPV group" will receive mask IPPV with an initial PIP of 20 cmH2O and PEEP of 5 cm H2O, and a ventilation rate of 40-60 inflations/min until spontaneously breathing, at which time CPAP will be provided.
  Arms: IPPV group
Procedure: SI group — Infants randomized into the "SI group" will receive two initial sustained inflations with a PIP of 20 cmH2O. After the two initial SIs infants will receive PEEP of 5 cm H2O and then CPAP if breathing spontaneously or, if found to have apnea or laboured breathing, mask IPPV with a PIP of 20 cmH2O and PEEP of 5 cmH2O at a rate of 40 to 60 bpm until spontaneously breathing, at which time CPAP will be provided
  Arms: "SI group"

SUMMARY:
To determine if respiratory support at birth guided by RFM decreases BPD.

DETAILED DESCRIPTION:
Despite recent advances in perinatal-neonatal care, there is an increasing trend of bronchopulmonary dysplasia (BPD) among survivors of prematurity1. Most infants developing BPD are born prematurely, and 75% of affected babies weigh less than 1000g at birth2. The risk of developing BPD increases with decreasing birth weight with reported incidence as high as 85% in neonates weighing between 500g and 699g, but only 5% in infants with birth weights over 1500g2. Alberta has the highest rate (10%) of delivering premature infants in Canada. In Edmonton approximately 200 premature infants <1250 g birth weight are born annually and up to 50% will develop BPD. This puts a heavy burden on health resources since these infants require frequent hospital re-admission in the first two years after birth and, even as adolescents have persistent respiratory symptoms.

Hypothesis Preterm infants <33 weeks gestation requiring breathing support at birth, the delivery of SIs (SI group) before mask ventilation compared to standard mask ventilation (IPPV group) will reduce the incidence of BPD.

Aim To determine if respiratory support at birth with initial sustained inflation compared to IPPV decreases BPD.

Study population Entry criteria Infants <33 weeks gestation born in the Royal Alexandra Hospital who require respiratory support for resuscitation in the delivery room.

Exclusion criteria Infants will be excluded if they have a congenital abnormality or condition that might have an adverse effect on breathing or ventilation, e.g. congenital pulmonary or airway anomalies, congenital diaphragmatic hernia, or congenital heart disease requiring intervention in neonatal period. Infants will also be excluded if their parents refuse to give consent to this study.

Description of interventions "SI group" Infants randomized into the "SI group" will receive two initial sustained inflations before PPV or CPAP.

"IPPV group" Infants randomized into the "IPPV group" will receive mask IPPV with an initial PIP of 20 cmH2O and PEEP of 5 cm H2O, and a ventilation rate of 40-60 inflations/min until spontaneously breathing, at which time CPAP will be provided.

"Failed SI or IPPV" Babies who fail to improve or remain apneic, bradycardic or hypoxemic despite two SIs and/or 30 seconds of effective IPPV require an alternative airway. Unit policy also dictates elective intubation and instillation of surfactant if, despite CPAP, a preterm infant continues to have increased work of breathing or requires a sustained inspiratory oxygen concentration over 40%.

ELIGIBILITY:
Inclusion Criteria:

* Infants <33 weeks gestation born in the Royal Alexandra Hospital who require respiratory support for resuscitation in the delivery room.

Exclusion Criteria:

* Infants will be excluded if they have a congenital abnormality or condition that might have an adverse effect on breathing or ventilation, e.g. congenital pulmonary or airway anomalies, congenital diaphragmatic hernia, or congenital heart disease requiring intervention in neonatal period. Infants will also be excluded if their parents refuse to give consent to this study.

Max Age: 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Difference in bronchopulmonary dysplasia | 36 weeks corrected gestational age
  Difference in bronchopulmonary dysplasia as defined by need for oxygen or respiratory support at 36 weeks corrected gestational age.

SECONDARY OUTCOMES:
Neonatal death < 28 days | < 28 days
  Neonatal death < 28 days
Death before discharge | before discharge from the NICU
  Death before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, MD,PhD, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Shah PS, Sankaran K, Aziz K, Allen AC, Seshia M, Ohlsson A, Lee SK; Canadian Neonatal Network. Outcomes of preterm infants <29 weeks gestation over 10-year period in Canada: a cause for concern? J Perinatol. 2012 Feb;32(2):132-8. doi: 10.1038/jp.2011.68. Epub 2011 May 19. PMID 21593814
- [Background] Baraldi E, Filippone M. Chronic lung disease after premature birth. N Engl J Med. 2007 Nov 8;357(19):1946-55. doi: 10.1056/NEJMra067279. No abstract available. PMID 17989387
- [Background] Kattwinkel J, Perlman JM, Aziz K, Colby C, Fairchild K, Gallagher J, Hazinski MF, Halamek LP, Kumar P, Little G, McGowan JE, Nightengale B, Ramirez MM, Ringer S, Simon WM, Weiner GM, Wyckoff M, Zaichkin J. Part 15: neonatal resuscitation: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S909-19. doi: 10.1161/CIRCULATIONAHA.110.971119. No abstract available. PMID 20956231
- [Background] Schmolzer GM, Te Pas AB, Davis PG, Morley CJ. Reducing lung injury during neonatal resuscitation of preterm infants. J Pediatr. 2008 Dec;153(6):741-5. doi: 10.1016/j.jpeds.2008.08.016. No abstract available. PMID 19014815
- [Background] Jobe AH. The New BPD. NeoReviews. 2006 Oct 1;7(10):e531-45.
- [Background] Boon AW, Milner AD, Hopkin IE. Lung expansion, tidal exchange, and formation of the functional residual capacity during resuscitation of asphyxiated neonates. J Pediatr. 1979 Dec;95(6):1031-6. doi: 10.1016/s0022-3476(79)80304-2. PMID 387935
- [Background] Vyas H, Milner AD, Hopkin IE, Boon AW. Physiologic responses to prolonged and slow-rise inflation in the resuscitation of the asphyxiated newborn infant. J Pediatr. 1981 Oct;99(4):635-9. doi: 10.1016/s0022-3476(81)80279-x. PMID 7277110
- [Background] Lindner W, Vossbeck S, Hummler H, Pohlandt F. Delivery room management of extremely low birth weight infants: spontaneous breathing or intubation? Pediatrics. 1999 May;103(5 Pt 1):961-7. doi: 10.1542/peds.103.5.961. PMID 10224173
- [Background] Lista G, Fontana P, Castoldi F, Cavigioli F, Dani C. Does sustained lung inflation at birth improve outcome of preterm infants at risk for respiratory distress syndrome? Neonatology. 2011;99(1):45-50. doi: 10.1159/000298312. Epub 2010 Jul 9. PMID 20616570
- [Background] te Pas AB, Walther FJ. A randomized, controlled trial of delivery-room respiratory management in very preterm infants. Pediatrics. 2007 Aug;120(2):322-9. doi: 10.1542/peds.2007-0114. PMID 17671058
- [Background] te Pas AB, Siew M, Wallace MJ, Kitchen MJ, Fouras A, Lewis RA, Yagi N, Uesugi K, Donath S, Davis PG, Morley CJ, Hooper SB. Effect of sustained inflation length on establishing functional residual capacity at birth in ventilated premature rabbits. Pediatr Res. 2009 Sep;66(3):295-300. doi: 10.1203/PDR.0b013e3181b1bca4. PMID 19542905
- [Background] Siew ML, Te Pas AB, Wallace MJ, Kitchen MJ, Lewis RA, Fouras A, Morley CJ, Davis PG, Yagi N, Uesugi K, Hooper SB. Positive end-expiratory pressure enhances development of a functional residual capacity in preterm rabbits ventilated from birth. J Appl Physiol (1985). 2009 May;106(5):1487-93. doi: 10.1152/japplphysiol.91591.2008. Epub 2009 Mar 26. PMID 19325025
- [Background] Schmolzer GM, Morley CJ, Wong C, Dawson JA, Kamlin CO, Donath SM, Hooper SB, Davis PG. Respiratory function monitor guidance of mask ventilation in the delivery room: a feasibility study. J Pediatr. 2012 Mar;160(3):377-381.e2. doi: 10.1016/j.jpeds.2011.09.017. Epub 2011 Nov 5. PMID 22056350
- [Background] Dawson JA, Schmolzer GM, Kamlin CO, Te Pas AB, O'Donnell CP, Donath SM, Davis PG, Morley CJ. Oxygenation with T-piece versus self-inflating bag for ventilation of extremely preterm infants at birth: a randomized controlled trial. J Pediatr. 2011 Jun;158(6):912-918.e1-2. doi: 10.1016/j.jpeds.2010.12.003. Epub 2011 Jan 15. PMID 21238983
- [Background] Dawson JA, Kamlin CO, Vento M, Wong C, Cole TJ, Donath SM, Davis PG, Morley CJ. Defining the reference range for oxygen saturation for infants after birth. Pediatrics. 2010 Jun;125(6):e1340-7. doi: 10.1542/peds.2009-1510. Epub 2010 May 3. PMID 20439604
- [Background] Rabi Y, Singhal N, Nettel-Aguirre A. Room-air versus oxygen administration for resuscitation of preterm infants: the ROAR study. Pediatrics. 2011 Aug;128(2):e374-81. doi: 10.1542/peds.2010-3130. Epub 2011 Jul 11. PMID 21746729
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Finer NN, Carlo WA, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Donovan EF, Newman NS, Ambalavanan N, Frantz ID 3rd, Buchter S, Sanchez PJ, Kennedy KA, Laroia N, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Bhandari V, Watterberg KL, Higgins RD. Early CPAP versus surfactant in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1970-9. doi: 10.1056/NEJMoa0911783. Epub 2010 May 16. PMID 20472939
- [Background] Morley CJ, Davis PG, Doyle LW, Brion LP, Hascoet JM, Carlin JB; COIN Trial Investigators. Nasal CPAP or intubation at birth for very preterm infants. N Engl J Med. 2008 Feb 14;358(7):700-8. doi: 10.1056/NEJMoa072788. PMID 18272893
- [Derived] Ngan AY, Cheung PY, Hudson-Mason A, O'Reilly M, van Os S, Kumar M, Aziz K, Schmolzer GM. Using exhaled CO2 to guide initial respiratory support at birth: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2017 Nov;102(6):F525-F531. doi: 10.1136/archdischild-2016-312286. Epub 2017 Jun 8. PMID 28596379